CLINICAL TRIAL: NCT04041427
Title: Development of Urinary-based Assay to Determine Treatment Coverage With Albendazole in Mass Drug Administration Programs
Brief Title: Urine Albendazole Levels for Coverage Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Salta (Other)
Collaborators: Fundacion Mundo Sano (Unknown); CIVETAN-Tandil, UNCPBA (Unknown); Natural History Museum, London, UK (Unknown)
Responsible Party: Principal Investigator, Alejandro Krolewiecki, Investigador CIC CONICET, Universidad Nacional de Salta
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ABZ0201
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Helminthiasis
MeSH Terms: conditions — Helminthiasis | interventions — Albendazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasting (Experimental): Albendazole 400mg will be ingested by study participants with an 8-hour fasting diet.
  Interventions: Drug: Albendazole Pill
- High fat content diet (Experimental): Albendazole 400mg will be ingested by study participants 15 to 30 minutes after a meal with high fat content (40 grams of fat).
  Interventions: Drug: Albendazole Pill; Other: High fat content diet
- Moderate fat content diet (Experimental): Albendazole 400mg will be ingested by study participants 15 to 30 minutes after a meal with moderate fat content (15 grams of fat).
  Interventions: Drug: Albendazole Pill; Other: Moderate fat content die

INTERVENTIONS:
Drug: Albendazole Pill — Albendazole 400mg po
Other: High fat content diet — High fat content diet
  Arms: High fat content diet
Other: Moderate fat content die — Moderate fat content die
  Arms: Moderate fat content diet

SUMMARY:
This project will develop and assess the feasibility and acceptability of a urine-based assay to monitor adherence to Mass Drug Administration (MDA) campaigns within Soil-transmitted helminthiasis (STH) control programs, evaluating the urine and serum pharmacokinetics of ALBENDAZOLE (ABZ) and its metabolites across a variety of food/fast conditions, age, gender and body weight. The final goal is to obtain a field ready tool for the measurement of adherence to anthelmintic treatment at a community level that serves as a coverage/adherence indicator and a reference standard for other monitoring tools.

DETAILED DESCRIPTION:
Soil-Transmitted-Helminthic (STH) infections are a major public health issue affecting the world's poorest populations. Control strategies for STH have been focused on the use of mass chemotherapy often delivered to school-aged-children; although there is strong interest in considering community wide MDA to achieve transmission interruption of STH. In these programs, directly observed treatment is not consistently or frequently achieved and so the verification of reported adherence is crucial to understanding of the impact of these programs.

It is important to differentiate a lack of adherence to treatment with albendazole (ABZ) from absorption/metabolism/resistance-related therapeutic failures. In that context, tools to evaluate, by means of non-invasive measures, treatment adherence either in adults or children, should be developed. In addition, drug absorption and metabolism among people may vary enormously depending on different factors such as genetics, age, gender, diet, weight and disease. Any of those factors may alter the ABZ/metabolites disposition kinetics and, consequently, the exposure of the target STH to the active drug.

The current research project proposes to establish evidence for the feasibility and usability of such a tool within MDA programs from the perspectives of the end-user (community), implementing partners, National Neglected Tropical Diseases (NTD) program and the World Health Organization. The proposed use case for this currently developed assay is to confirm the findings of the standard coverage survey (based on self-report) in the context of community MDA. Further validation and technical development of a field ready tool for monitoring adherence to albendazole, in addition to the identification of key factors affecting drug therapeutic response is proposed within this project.

Main goals of the current proposal:

1. To assess key factors affecting the feasibility of using a urinary assay to monitor adherence to MDA within STH control programs, including tool acceptability, tool learnability, system capacity to deliver, timing of administration, frequency of administration, adequate breadth of administration, sustainability of use, responsiveness of health systems to tool output, and efficiency of administration.
2. To evaluate the influence of diet, fasting, age, gender and body weight on the serum disposition kinetics and pattern of urinary excretion of ABZ/metabolites in non-infected human volunteers.
3. To evaluate the relationship between drug serum/urine concentrations with potential factors affecting ABZ/metabolites disposition kinetics in children.
4. To characterize the pattern of amino-ABZSO2 urinary excretion in non-infected human volunteers treated with ABZ and to determine the longest period of time after ABZ treatment where amino-ABZSO2 can be measured in urine (alternatively to ABZSO) as an indirect assessment of an individual's adherence to treatment.
5. To determine drug/metabolites chemical stability in urine samples at different temperatures (reproducing environmental conditions of tropical weather).

Study procedures:

Twelve (12) healthy adult volunteers (body weight between 45 and 75 kg, women n=6 and men n=6) will participate in a crossover design with three (3) different experimental phases. In Phase I, volunteers will be assigned to either Group I, Group II or Group III (n=4 each, two female and two male individuals). In the following 2 Phases of the study, volunteers will be cross-over between the other 2 Groups, with a 14-day washout period between Phases. All groups and phases will receive 400 mg of ABZ (Glaxo SmithKline).

Group I (heavy meal):30 minutes after a high-fatty meal (estimated fat content 40 g).

Group II (light meal):30 minutes after a light meal (infusion tea). Group III (fasted):at 8-hours fasting condition.

Prior to ABZ treatment (sampling time =0), a baseline blood (5 mL) and urine (10 mL) samples will be obtained in each phase. Venous blood samples will be collected at 2, 4, 8, 12, 24, 36, 48 and 72 h, after ABZ administration. Urine samples will be collected at 2, 4, 8, 12, 24, 36, 48 and 72 h post-treatment. Samples will be stored at -20ºC until HPLC analysis of ABZ/metabolites.

Urine samples from time 4-hours will be aliquoted in 3 in order to evaluate the effect of storage at 32°C (in an incubator) for 12 and 24 hours before freezing at -20°C in the measurement of drug/metabolite levels. A total of 12 samples from Group 1 will be included in this sub-sample analysis which will provide information on the stability of the samples at temperatures in tropical environments.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: 18 to 25.
* Physical exam without significant abnormal findings

Exclusion Criteria:

* Pregnancy
* Lactation
* Use of ABZ or other benzimidazole drugs in the previous 30 days.
* History of intolerance to ABZ.
* Malabsorption and/or other gastrointestinal conditions that might compromise ABZ absorption.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Urine albendazole levels | 96 hours
  Albendazole and its metabolites will be measured in urine samples through high performance liquid chromatography (HPLC).
Serum albendazole levels | 72 hours
  Albendazole and its metabolites will be measured in serum samples obtained from venous blood through HPLC.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Investigaciones de Enfermedades Tropicales, UNSalta, Orán, Salta Province, Argentina

IPD SHARING:
Plan to Share IPD: No